CLINICAL TRIAL: NCT00450008
Title: Phase II Study of Patients With Hormone-Naïve Prostate Cancer With a Rising Prostate Specific Antigen: Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF), Thalidomide Plus Docetaxel
Brief Title: Safety and Efficacy Study of GM-CSF, Thalidomide Plus Docetaxel in Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI decision
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMRI IRB#1006-0153; PCa-06-102 (Other: Principal Investigator)
Record Dates: First submitted 2007-03-19; First posted 2007-03-21 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate Cancer; Hormone-Naïve Prostate Cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Thalidomide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): Combination therapy of GM-CSF, Thalidomide plus Docetaxel in patients with prostate cancer with a rising PSA
  Interventions: Drug: GM-CSF; Drug: thalidomide; Drug: docetaxel

INTERVENTIONS:
Drug: GM-CSF — fixed dose of 250 mcg/m2, 3 days per week by subcutaneous injection
  Other Names: Leukine
Drug: thalidomide — Thalidomide by oral administration at a fixed dose of 200 mg. Prophylactic Coumadin® by oral administration at a fixed dose of 2.5 mg to prevent thromboembolic events (DVT and TIA/stroke) during Thalidomide administration. Thalidomide and Coumadin will be given daily at bedtime without interruption.
  Other Names: Thalomid
Drug: docetaxel — Docetaxel will be administered by intravenous piggyback over 1 hour at 75mg/m² every 3 weeks. Pre-medication for the docetaxel infusion will consist of dexamethasone 8 mg administered orally 12 hours, 3 hours and 1 hour before docetaxel.
  Other Names: Taxotere

SUMMARY:
The purpose of this study is to assess the relative efficacy and toxicity of combination therapy of GM-CSF, Thalidomide plus Docetaxel in patients with prostate cancer with a rising PSA.

DETAILED DESCRIPTION:
As more men are being diagnosed and treated for prostate cancer at an early age, the number who experiences a rising level of prostate-specific antigen (PSA) after initial treatment is increasing, affecting approximately 50,000 patients each year.

These three drugs are commercially available. Thalidomide is an angiogenesis inhibitor which blocks the development of new blood vessels. GM-CSF stimulates the body's immune response to fight cancer. Docetaxel is the most active chemotherapeutic agent in the treatment of prostate cancer. GM-CSF and thalidomide have proven activity in suppressing PSA values.

This study design offers an opportunity to add cytotoxic therapy (docetaxel) in combination with an active pathobiologic regimen (GM-CSF plus thalidomide) to eradicate micrometastatic disease, thus potentially offering a significant delay to clinical failure as measured by a rise in PSA or radiographic involvement. Additionally, delays in the use of hormone therapy has the potential to be of significant benefit.

GM-CSF will be administered at a fixed dose 3 days per week by subcutaneous injection for 12 months. Participants will receive a fixed dose of thalidomide orally at bedtime daily without interruption for 12 months. Docetaxel will be administered intravenously over 1 hour on week 1 of every cycle (every 3 weeks) for 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adenocarcinoma of the prostate.
* Failure of local treatments (surgery and/or radiation) as defined by a rising PSA; demonstrated by at least three consecutive rises in PSA by intervals of at least 4 weeks apart with an absolute change of at least 1 ng/mL. If the confirmatory PSA (third PSA) is less than the previous screening PSA value, an additional test for rising PSA will be required to document progression.
* No clinical or radiographic evidence of disease.
* The Zubrod performance status 0-1.
* Prior hormonal therapy in the form of neoadjuvant or adjuvant therapy is allowed as long as androgen therapy has been completed at least 1 year prior to study entry.
* Adequate hematologic function: absolute granulocytes ≥ 1500/ul, platelets ≥ 100,000/ul, hemoglobin ≥ 10 gm/100 ml within 4 weeks prior to study entry.
* Adequate hepatic function: bilirubin ≤ 1.5 mg/dl, liver enzymes ≤ 1.5 ULN within 4 weeks prior to study entry.
* Adequate renal function: creatinine ≤ 1.5 x ULN within 4 weeks prior to study entry.
* Patients treated with bisphosphonate therapy before or after study entry are eligible to continue in the study.
* Negative bone scan within 6 weeks prior to study entry.
* Negative CT scan or MRI of the abdomen and pelvis within 6 weeks prior to study entry.
* Negative chest x-ray for metastatic disease within 6 weeks prior to study entry.
* Patients must sign a written informed consent prior to treatment.

Exclusion Criteria:

* Serious intercurrent medical illness including symptomatic heart disease within 6 months.
* Previous or concurrent invasive cancers other than superficial non-melanomatous skin cancer unless disease-free for at least 5 years.
* Major medical or psychiatric illness which, in the investigator's opinion, would prevent completion of treatment and would interfere with follow-up.
* History of thromboembolic events (deep venous thrombosis, symptomatic cerebrovascular events or pulmonary embolism), history of MI, within the last 12 months.
* History of bleeding disorders that would contraindicate Coumadin® (warfarin) including: esophageal varices and clotting factor defects

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-12; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To assess the relative efficacy of the combination of GM-CSF, Thalidomide and Docetaxel in patients with prostate cancer. | during study (no data currently available)
  PI relocated, no data currently available

SECONDARY OUTCOMES:
Collect data on hormonal responses produced by GM-CSF, Thalidomide and Docetaxel. | during study (no data currently available)
  PI relocated, no data currently available
Evaluate safety and toxicity of the combination of GM-CSF, Thalidomide and Docetaxel for patients with hormone naïve prostate cancer. | during study (no data currently available)
  PI relocated, no data currently available

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, DO, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- The Methodist Hospital Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No